CLINICAL TRIAL: NCT00012441
Title: Comparison of Daily Nocturnal Hemodialysis With Daily Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0781
Record Dates: First submitted 2001-03-06; First posted 2001-03-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Failure, Chronic
Keywords: Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

INTERVENTIONS:
Procedure: hemodialysis

SUMMARY:
Hemodialysis remains associated with a high mortality (approximately 22% per year) and many complications despite improvements over the last twenty years. Several nephrologists have suggested that increasing the frequency and amount of dialysis will result in improved outcomes. In fact, various forms of daily dialysis have been performed in over 300 patients in the last 30 years with improvements in blood pressure, quality-of-life, bone disease, and other complications of renal failure. Whether this form of treatment can be expanded to the 220,000 Americans on hemodialysis is unknown. The primary outcome of this study is to determine the effectiveness of nocturnal dialysis in hemodialysis patients in St. Louis. If the pilot study is effective, then participation in a larger, multicenter trial is expected. The endpoints measured are use of antihypertensive medications, improvement in secondary hyperparathyroidism and use of phosphorus binders, quality-of-life measured by SF-36 surveys, and improvement in physical function as measured by maximal oxygen uptake.

ELIGIBILITY:
Adult patients with chronic renal failure requiring intermittent hemodialysis with a life expectancy of greater than 2 years

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States